CLINICAL TRIAL: NCT07205471
Title: The Clinical Efficacy of Laparoscopic Partial Splenectomy for Hypersplenism in Liver Cirrhosis Patients
Brief Title: Laparoscopic Partial Splenectomy for Hypersplenism in Liver Cirrhosis Patients
Acronym: LPSH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Guo-Qing Jiang, Clinical Professor, Northern Jiangsu People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YZUC-014
Record Dates: First submitted 2025-09-14; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Cirrhoses, Liver; Splenectomy; Status; Partial
Keywords: Cirrhosis; Splenectomy; Laparoscopy; immune function; partial
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic splenectomy (No Intervention): Patients in this arm undergo the standard laparoscopic splenectomy procedure, which serves as the active comparator. The entire spleen is removed after careful dissection and ligation of the splenic hilum.
- laparoscopic partial splenectomy (Experimental): The laparoscopic partial splenectomy technique involved preserving the short gastric vessels and the splenic suspensory ligament, with resection conducted along the demarcation line.
  Interventions: Procedure: Laparoscopic Partial Splenectomy

INTERVENTIONS:
Procedure: Laparoscopic Partial Splenectomy — The laparoscopic partial splenectomy technique involved preserving the short gastric vessels and the splenic suspensory ligament, with resection conducted along the demarcation line.
  Arms: laparoscopic partial splenectomy

SUMMARY:
In this study,the researchers compared the changes in immune function-related indicators in patients with liver cirrhosis following laparoscopic partial splenectomy,to determine whether this surgical intervention can enhance postoperative immune function and thereby improve patient outcomes.

DETAILED DESCRIPTION:
Patients meeting the study's inclusion criteria were enrolled, and their baseline demographic data were collected. Eligible patients were randomly assigned in a 1:1 ratio to two groups: the laparoscopic splenectomy group and the laparoscopic partial splenectomy group, using a computer-generated randomization sequence. Following comprehensive preoperative preparation, all surgeries were performed by the same surgical team. The laparoscopic partial splenectomy technique involved preserving the short gastric vessels and the splenic suspensory ligament, with resection conducted along the demarcation line.

Postoperatively, all patients received standardized care from the same nursing team, followed by a uniform treatment protocol that included pharmacotherapy, additional therapeutic interventions, and follow-up assessments. Throughout the treatment period, monitoring was performed preoperatively and at 7 days, 1, 3, 6, and 12 months postoperatively. The parameters monitored included routine blood tests, liver function, coagulation profile, immune function, and hemodynamics of the portal vein, proper hepatic artery, and splenic vein.Additionally, indocyanine green (ICG) clearance tests were performed at 3, 6, and 12 months to assess liver function.

ELIGIBILITY:
Inclusion Criteria:

* A clinical, radiological or histologic diagnosis of cirrhosis of any etiology
* Splenomegaly with secondary hypersplenism
* gastroesophageal variceal bleeding
* Informed consent to participate in the study

Exclusion Criteria:

* Hepatocellular carcinoma or any other malignancy,
* Child-Pugh grade C
* Recent peptic ulcer disease
* History of Hemorrhagic stroke
* Pregnancy.
* Uncontrolled Hypertension
* Human immunodeficiency virus (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2028-09-24 (Estimated); Study Completion 2028-09-24 (Estimated)

PRIMARY OUTCOMES:
Change in Humoral Immune Markers from Baseline to 6 Months Postoperation | Baseline (preoperative) and 6 months postoperation
  Serum levels of immunoglobulins (IgG, IgA, IgM), complement proteins (C3, C4), and B-cell markers (CD19, CD20) will be measured. The primary outcome is the change in these markers from preoperative baseline to 6 months after surgery.
Platelet Count at 6 Months Postoperation | 6 months postoperation
  Platelet count (×10⁹/L) will be measured and compared between the two surgical groups.
White Blood Cell Count at 6 Months Postoperation | 6 months postoperation
  White blood cell count (×10⁹/L) will be compared between groups.
Hemoglobin Level at 6 Months Postoperation | 6 months postoperation
  Hemoglobin concentration (g/L) will be compared between groups.
Blood Flow Velocity of the Portal Vein at 6 Months Postoperation | 6 months postoperation
  Blood flow velocity (cm/s) in the portal vein, measured by Doppler ultrasound, will be compared between groups.
Vascular Diameter of the Portal Vein at 6 Months Postoperation | 6 months postoperation
  Vascular diameter (mm) of the portal vein, measured by Doppler ultrasound, will be compared between groups.
Blood Flow Velocity of the Splenic Vein at 6 Months Postoperation | 6 months postoperation
  Blood flow velocity (cm/s) in the splenic vein, measured by Doppler ultrasound, will be compared between groups.
Vascular Diameter of the Splenic Vein at 6 Months Postoperation | 6 months postoperation
  Vascular diameter (mm) of the splenic vein, measured by Doppler ultrasound, will be compared between groups.
Indocyanine Green Retention Rate at 15 Minutes (ICG R15) at 6 Months Postoperation | 6 months postoperation
  Indocyanine green retention rate at 15 minutes (%), a measure of liver function, will be compared between groups.
Incidence of Portal Venous System Thrombosis within 6 Months Postoperation | 6 months postoperation
  The number of participants with newly developed thrombosis in the portal venous system, confirmed by imaging, will be recorded and compared.

SECONDARY OUTCOMES:
Comparison of Humoral Immune Marker Levels at 7 Days Postoperation | 7 days postoperation
  Serum levels of key humoral immune markers (including but not limited to IgG, IgA, IgM, C3, C4, CD19, CD20) will be compared between the laparoscopic partial splenectomy group and the total splenectomy group at 7 days after surgery.
Comparison of Humoral Immune Marker Levels at 3 months Postoperation | 3 months postoperation
  Serum levels of key humoral immune markers (IgG, IgA, IgM, C3, C4, CD19, CD20) will be compared between the two groups at this time point
Platelet Count at 3 Months Postoperation | 3 months postoperation
  Platelet count (×10⁹/L) will be measured and compared between the two surgical groups.
Platelet Count at 12 Months Postoperation | 12 months postoperation
  Platelet count (×10⁹/L) will be measured and compared between the two surgical groups.
Platelet Count at 1 Month Postoperation | 1 month postoperation
  Platelet count (×10⁹/L) will be measured and compared between the two surgical groups.
Comparison of Humoral Immune Marker Levels at 1 Month Postoperation | 1 month postoperation
  Serum levels of key humoral immune markers (IgG, IgA, IgM, C3, C4, CD19, CD20) will be compared between the two groups at this time point.
Comparison of Humoral Immune Marker Levels at 12 Months Postoperation | 12 Months postoperation
  Serum levels of key cellular immune markers (CD4, CD16, CD56, CD35) will be compared between the two groups at this time point.
White Blood Cell Count at 1 Month Postoperation | 1 month postoperation
  White blood cell count (×10⁹/L) will be compared between groups.
White Blood Cell Count at 3 Months Postoperation | 3 months postoperation
  White blood cell count (×10⁹/L) will be compared between groups
White Blood Cell Count at 12 Months Postoperation | 12 months postoperation
  White blood cell count (×10⁹/L) will be compared between groups.
Hemoglobin Level at 1 Month Postoperation | 1 month postoperation
  Hemoglobin concentration (g/L) will be compared between groups.
Hemoglobin Level at 3 Months Postoperation | 3 months postoperation
  Hemoglobin concentration (g/L) will be compared between groups.
Hemoglobin Level at 12 Months Postoperation | 12 months postoperation
  Hemoglobin concentration (g/L) will be compared between groups.
Blood Flow Velocity of the Portal Vein at 3 Months Postoperation | 3 months postoperation
  Blood flow velocity (cm/s) in the portal vein, measured by Doppler ultrasound, will be compared between groups.
Blood Flow Velocity of the Portal Vein at 12 Months Postoperation | 12 months postoperation
  Blood flow velocity (cm/s) in the portal vein, measured by Doppler ultrasound, will be compared between groups.
Vascular Diameter of the Portal Vein at 3 Months Postoperation | 3 months postoperation
  Vascular diameter (mm) of the portal vein, measured by Doppler ultrasound, will be compared between groups.
Vascular Diameter of the Portal Vein at 12 Months Postoperation | 12 months postoperation
  Vascular diameter (mm) of the portal vein, measured by Doppler ultrasound, will be compared between groups.
Blood Flow Velocity of the Splenic Vein at 3 Months Postoperation | 3 months postoperation
  Blood flow velocity (cm/s) in the splenic vein, measured by Doppler ultrasound, will be compared between groups.
Blood Flow Velocity of the Splenic Vein at 12 Months Postoperation | 12 months postoperation
  Blood flow velocity (cm/s) in the splenic vein, measured by Doppler ultrasound, will be compared between groups.
Vascular Diameter of the Splenic Vein at 3 Months Postoperation | 3 months postoperation
  Vascular diameter (mm) of the splenic vein, measured by Doppler ultrasound, will be compared between groups.
Vascular Diameter of the Splenic Vein at 12 Months Postoperation | 12 months postoperation
  Vascular diameter (mm) of the splenic vein, measured by Doppler ultrasound, will be compared between groups.
Indocyanine Green Retention Rate at 15 Minutes (ICG R15) at 3 Months Postoperation | 3 months postoperation
  Indocyanine green retention rate at 15 minutes (%), a measure of liver function, will be compared between groups.
Indocyanine Green Retention Rate at 15 Minutes (ICG R15) at 9 Months Postoperation | 9 months postoperation
  Indocyanine green retention rate at 15 minutes (%), a measure of liver function, will be compared between groups.
Indocyanine Green Retention Rate at 15 Minutes (ICG R15) at 12 Months Postoperation | 12 months postoperation
  Indocyanine green retention rate at 15 minutes (%), a measure of liver function, will be compared between groups.
Incidence of Portal Venous System Thrombosis within 12 Months Postoperation | 12 months postoperation
  The number of participants with newly developed thrombosis in the portal venous system, confirmed by imaging, will be recorded and compared.
Incidence of Postoperative Complications within 30 Days | 30 days postoperation
  The number of participants experiencing complications (e.g., bleeding, infection, pancreatic fistula) will be compared using the Clavien-Dindo classification or similar.

CONTACTS AND LOCATIONS:
Overall Officials: Guo-Qing Jiang, Study Chair — Clinical Medical College, Yangzhou University
Locations (1):
- Clinical Medical College of Yangzhou University, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No